CLINICAL TRIAL: NCT02839005
Title: Absorbable Suture Versus Nonabsorbable Suture Intradermal for the Skin Transverse Section in Cesarean
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade do Vale do Sapucai (Other)
Responsible Party: Principal Investigator, Roberta Junqueira Lima, MD, Universidade do Vale do Sapucai
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: MRJ
Record Dates: First submitted 2016-07-18; First posted 2016-07-20 (Estimated); Last update posted 2016-07-20 (Estimated); Status verified 2016-07

CONDITIONS: Cesarean Section; Sutures
Keywords: Wound Closure Thechnical; Wound Healing
MeSH Terms: interventions — glycolide E-caprolactone copolymer; Nylons

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- suture with polyglecaprone 25 (Active Comparator)
  Interventions: Other: Continuous suture with polyglecaprone 25
- suture with polyamide (nylon) (Active Comparator)
  Interventions: Other: Continuous suture with polyamide (nylon)

INTERVENTIONS:
Other: Continuous suture with polyglecaprone 25 — At the end of surgical procedemento of cesarean delivery , for skin closure continuous suture was performed with polyglecaprone 25
  Arms: suture with polyglecaprone 25
Other: Continuous suture with polyamide (nylon) — At the end of surgical procedemento of cesarean delivery , for skin closure continuous suture was performed with polyamide (nylon)
  Arms: suture with polyamide (nylon)

SUMMARY:
Context: Cesarean section is the most common surgery in women, both in developed and underdeveloped countries. However results are conflicting report in which material for intradermal suturing get better aesthetic result. Objective: To compare the aesthetic appearance of two suture materials, polyglecaprone 25 and polyamide (nylon) with intradermal sutures for skin closure in women undergoing cesarean section first. Methods: This is a clinical, prospective and randomized study which was conducted in the Department of Gynecology and Obstetrics of a tertiary Institute, Hospital das Clinicas Samuel Libânio, in PousoAlegre, Estate of Minas Gerais. Sixty women undergoing cesarean section were first included and randomized into two groups: group I (n = 30) polyamide and group II (n = 30) polyglecaprone 25. Hypertrophy, color and width of the wound were evaluated, receiving a score, according to Trimbos table, six months after surgery. Later the results were compared to non-parametric statistical tests

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent cesarean section
* No restriction of ethnicity, education or social class

Exclusion Criteria:

* Scarring Pfannenstiel prior
* Diabetic patients using drugs;
* Patients with collagen diseases
* Patients with pre operative tests to indicate any systemic sign of infection or site, not previously treated until the time of surgery.
* Patients who withdrew informed consent
* Patients who did not attend the pre scheduled dates for the controls after surgery .

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-04; Primary Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Photographic documentation for evaluation | 6 Months
  The photographic record was sent to three experts for evaluation of hypertrophy and cross marks staining points, according Trimboset al.,1993
Photographic documentation for evaluation | 6 Months
  The photographic record was sent to another expert for evaluation of hypertrophy and cross marks staining points, according Trimboset al.,1993, besides scar mesure

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital das Clínicas Samuel Libânio, Pouso Alegre, Minas Gerais, Brazil